CLINICAL TRIAL: NCT02454608
Title: Randomized Double Blind Placebo Controlled Trial of Verapamil in Chronic Rhinosinusitis
Brief Title: Trial of Verapamil in Chronic Rhinosinusitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Evidence that the dose is insufficient.
Sponsor: Benjamin Bleier (Other)
Responsible Party: Sponsor-Investigator, Benjamin Bleier, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-009H
Record Dates: First submitted 2015-05-11; First posted 2015-05-27 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Sinusitis; Nasal Polyps
MeSH Terms: conditions — Sinusitis; Nasal Polyps | interventions — Verapamil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment (Experimental): Verapamil HCl, capsules for oral administration, 80mg, TID, for 8 weeks
  Interventions: Drug: Verapamil HCl
- Control (Placebo Comparator): Placebo, capsules for oral administration, TID, for 8 weeks
  Interventions: Other: Placebo
- Open Label (Experimental): Verapamil HCl, capsules for oral administration, 80mg, TID, for 1 year
  Interventions: Drug: Verapamil HCl

INTERVENTIONS:
Drug: Verapamil HCl — Verapamil represents a calcium channel blocker which binds to the alpha subunit of L-type voltage dependent calcium (Cav1) channels thereby blocking the influx of calcium ions into the host cell. While Verapamil is classically used to promote the relaxation of cardiac and smooth muscle cells, recent evidence has suggested that it may also function as an immunomodulator in astrocytes, hepatocytes, and T-cells. Further research has demonstrated that Verapamil is capable of specifically reducing Th2 associated inflammation in asthma. These findings raise the provocative question as to whether Verapamil could also be effective in reducing inflammation in chronic rhinosinusitis with nasal polyps.
  Other Names: Verapamil
  Arms: Open Label; Treatment
Other: Placebo — Capsule with the same characteristics (size, color, smell) as Verapamil HCl.
  Arms: Control

SUMMARY:
Verapamil is an L-type calcium channel blocker(CCB) which has been shown to reduce inflammation in a variety of tissues. Verapamil has also been shown to improve eosinophilic inflammation in an animal model of asthma and also functions as a P-glycoprotein(P-gp) inhibitor. A major subtype of chronic rhinosinusitis(CRS) is characterized by eosinophilic inflammation as well as P-gp overexpression. The goal of this study is to therefore see whether Verapamil may be used to treat CRS.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) impacts more than 30 million Americans resulting in $6.9 to $9.9 billion in annual healthcare expenditures and $12.8 billion in productivity costs. The prevalence of Chronic Rhinosinusitis with Nasal Polyps(CRSwNP) in Europe has been estimated to be 2-4.3% and is thought to be similar in the United States. Corticosteroids remain the mainstay of treatment although novel therapies are being developed based on an evolving understanding of the inflammatory pathways involved in disease pathogenesis. CRSwNP is characterized by the presence of edematous polypoid mucosa and predominantly eosinophilic inflammation. Recent evidence has focused on the sinonasal epithelial cell as a primary driver of the local dysregulated immune response through secretion of type 2 helper T-cell(Th2) promoting cytokines. While these studies suggest that epithelial cells are capable of orchestrating a local immune response, the mechanisms responsible for regulating cytokine secretion are poorly understood and may be influenced by the efflux function of epithelial P-glycoprotein(P-gp).

P-gp is a 170 kiloDalton membrane protein which belongs to sub-family B of the adenosine triphosphate(ATP)-binding cassette(ABC) transporter superfamily. P-gp utilizes ATP hydrolysis to transport a wide range of substrates across the plasma membrane. P-gp mediated transport has been observed in the regulation of cytokine secretion in both human T-cells as well as sinonasal epithelial cells implicating a potential immunomodulatory role. Studies by our group have demonstrated that P-gp is overexpressed in the mucosa of patients with Th2 skewed CRS endotypes including CRSwNP and is capable of regulating the secretion of Th2 polarizing cytokines. Together, these findings suggest that P-gp participates in the non-canonical regulation of cytokine secretion within CRSwNP and may thereby represent a druggable target.

Verapamil Hydrochloride(HCl) was one of the first inhibitors of P-gp to be identified in 1982 and also functions as a calcium channel blocker(CCB). Verapamil has since been categorized as a first generation P-gp inhibitor as more potent and selective 2nd and 3rd generation molecules were subsequently developed for use as chemotherapy sensitizers. Several studies, including those by our group, have reported that Verapamil is capable of modulating inflammatory responses in human T-cells, animal models of asthma, and nasal polyps. Using an organotypic explant model, we have previously shown that Verapamil has similar effects to dexamethasone in its ability to abrogate Interleukin(IL)-5, IL-6, and Thymic Stromal Lymphopoietin secretion. While Verapamil is cardioactive, it is considered the first-line prophylactic drug for cluster headache and is usually well tolerated by otherwise healthy patients.

In light of our prior studies demonstrating the immunomodulatory role of P-gp in promoting Th2 skewing cytokine secretion in CRSwNP, we hypothesized that low dose Verapamil HCl monotherapy would be safe and effective in the treatment of CRSwNP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to the Massachusetts Eye and Ear Sinus Center
2. Age 18-80 yrs old
3. Diagnosed with Chronic Rhinosinusitis with Nasal Polyps according to the EPOS 2012 consensus criteria

Exclusion Criteria:

1. Patients with the following comorbidities:

   * GI Hypomotility
   * Heart Failure
   * Liver Failure
   * Kidney Disease
   * Muscular Dystrophy
   * Pregnant or Nursing Females
   * Steroid Dependency
2. Patients taking the following medications:

   * Aspirin
   * Beta-blockers
   * Cimetidine(Tagamet)
   * Clarithromycin(Biaxin)
   * Cyclosporin
   * Digoxin
   * Disopyramide(Norpace)
   * Diuretics
   * Erythromycin
   * Flecainide
   * HIV Protease Inhibitors(Indinavir, Nelfinavir, Ritonavir)
   * Quinidine
   * Lithium
   * Pioglitazone
   * Rifampin
   * St Johns Wort
3. Patients with cardiac or conduction abnormality picked up by screening EKG

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Bleier, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin D, Harvey RJ. Nasal polyposis: an inflammatory condition requiring effective anti-inflammatory treatment. Curr Opin Otolaryngol Head Neck Surg. 2013 Feb;21(1):23-30. doi: 10.1097/MOO.0b013e32835bc3f9. PMID 23172039
- [Background] Poetker DM, Jakubowski LA, Lal D, Hwang PH, Wright ED, Smith TL. Oral corticosteroids in the management of adult chronic rhinosinusitis with and without nasal polyps: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2013 Feb;3(2):104-20. doi: 10.1002/alr.21072. Epub 2012 Aug 7. PMID 22887970
- [Background] Khakzad MR, Mirsadraee M, Mohammadpour A, Ghafarzadegan K, Hadi R, Saghari M, Meshkat M. Effect of verapamil on bronchial goblet cells of asthma: an experimental study on sensitized animals. Pulm Pharmacol Ther. 2012 Apr;25(2):163-8. doi: 10.1016/j.pupt.2011.11.001. Epub 2011 Nov 25. PMID 22133887
- [Background] Matsumori A, Nishio R, Nose Y. Calcium channel blockers differentially modulate cytokine production by peripheral blood mononuclear cells. Circ J. 2010 Mar;74(3):567-71. doi: 10.1253/circj.cj-09-0467. Epub 2010 Jan 30. PMID 20118567
- [Background] Hashioka S, Klegeris A, McGeer PL. Inhibition of human astrocyte and microglia neurotoxicity by calcium channel blockers. Neuropharmacology. 2012 Sep;63(4):685-91. doi: 10.1016/j.neuropharm.2012.05.033. Epub 2012 May 30. PMID 22659089
- [Background] Li G, Qi XP, Wu XY, Liu FK, Xu Z, Chen C, Yang XD, Sun Z, Li JS. Verapamil modulates LPS-induced cytokine production via inhibition of NF-kappa B activation in the liver. Inflamm Res. 2006 Mar;55(3):108-13. doi: 10.1007/s00011-005-0060-y. PMID 16673153
- [Background] Bacon KB, Westwick J, Camp RD. Potent and specific inhibition of IL-8-, IL-1 alpha- and IL-1 beta-induced in vitro human lymphocyte migration by calcium channel antagonists. Biochem Biophys Res Commun. 1989 Nov 30;165(1):349-54. doi: 10.1016/0006-291x(89)91076-0. PMID 2686646
- [Background] Becker WJ. Cluster headache: conventional pharmacological management. Headache. 2013 Jul-Aug;53(7):1191-6. doi: 10.1111/head.12145. Epub 2013 Jun 14. PMID 23773141
- [Background] Cohen AS, Matharu MS, Goadsby PJ. Electrocardiographic abnormalities in patients with cluster headache on verapamil therapy. Neurology. 2007 Aug 14;69(7):668-75. doi: 10.1212/01.wnl.0000267319.18123.d3. PMID 17698788
- [Background] Lanteri-Minet M, Silhol F, Piano V, Donnet A. Cardiac safety in cluster headache patients using the very high dose of verapamil (>/=720 mg/day). J Headache Pain. 2011 Apr;12(2):173-6. doi: 10.1007/s10194-010-0289-x. Epub 2011 Jan 22. PMID 21258839
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl. 2012 Mar;23:3 p preceding table of contents, 1-298. PMID 22764607
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277

RESULTS

PARTICIPANT FLOW:
Period: Double-Blind Period
Arm/Group | Treatment | Control | Open Label
Started | 15 | 14 | 0 (This arm is not part of this period of the study)
Completed | 15 | 12 | 0 (This arm is not part of this period of the study)
Not Completed | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0
Period: Open Label Period
Arm/Group | Treatment | Control | Open Label
Started | 0 (This arm is not part of this period of the study) | 0 (This arm is not part of this period of the study) | 29
Completed | 0 (This arm is not part of this period of the study) | 0 (This arm is not part of this period of the study) | 10
Not Completed | 0 | 0 | 19
Not completed — Lost to Follow-up | 0 | 0 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Population: Intention-to-treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Open Label | Total
Number analyzed (Participants) | 10 | 10 | 29 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (14.7) | 48.4 (11.3) | 47.8 (11.7) | 48.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 10 | 18
  Male | 6 | 6 | 19 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4
  White | 7 | 8 | 24 | 39
  More than one race | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 29 | 49

OUTCOME MEASURES:

1. Primary Outcome: Subjective Sinonasal Symptoms on Sinonasal Outcomes Test-22(SNOT-22)
Description: Minimum Score: 0 Maximum Score: 110 A higher score indicates a worse outcome
Time Frame: baseline to week 8
Population: Intention-to-treat analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 10 | 10
units on a scale | -27.3 (7.52) | 0.4 (7.52)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

2. Primary Outcome: Subjective Sinonasal Symptoms on 10cm Visual Analogue Scale(VAS)
Description: Minimum Score: 0 Maximum Score: 100 A higher score indicates a worse outcome.
Time Frame: baseline to week 8
Population: Intention-to-treat analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 10 | 10
units on a scale | -44.03 (7.66) | -6.07 (7.66)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

3. Secondary Outcome: Objective Sinonasal Symptoms on Lund-Kennedy Score(LKS)
Description: Minimum Score: 0 Maximum Score: 12 Higher value represents worse outcome.
Time Frame: baseline to week 8
Population: Intention-to-treat analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 10 | 10
units on a scale | -1.3 (0.63) | -0.25 (0.63)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.25, Mixed Models Analysis

4. Secondary Outcome: Objective Sinonasal Symptoms on Lund-McKay Score(LMS)
Description: Minimum Score: 0 Maximum Score: 24 Higher value represents worse outcome.
Time Frame: Week 8
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 12.5 (4.4) | 17.7 (4.9)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

5. Other Pre Specified Outcome: Heart Rate
Time Frame: Mean change between baseline and week 8 measurements.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Treatment | Control
Number analyzed (Participants) | 10 | 10
beats per minute | -1.4 (9.16) | 4 (30.37)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.6, t-test, 2 sided

6. Other Pre Specified Outcome: Systolic Blood Pressure
Time Frame: Mean change between baseline and week 8 measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment | Control
Number analyzed (Participants) | 10 | 10
mmHg | -4.5 (13.2) | -6.6 (19.48)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.78, t-test, 2 sided

7. Other Pre Specified Outcome: Diastolic Blood Pressure
Time Frame: Mean change between baseline and week 8 measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment | Control
Number analyzed (Participants) | 10 | 10
mmHg | -0.6 (10.26) | 1 (7.85)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.7, t-test, 2 sided

8. Primary Outcome: Subjective Sinonasal Symptoms on Sinonasal Outcomes Test-22(SNOT-22)
Description: Minimum Score: 0 Maximum Score: 110 A higher score indicates a worse outcome
Time Frame: baseline to week 56
Population: Intention-to-treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 29
units on a scale
  Medicine Completers, baseline: number analyzed (Participants) | 7
  Medicine Completers, baseline | 31.8 (5.24)
  Medicine Completers, week 56: number analyzed (Participants) | 7
  Medicine Completers, week 56 | 24.14 (6.17)
  Surgical Completers, baseline: number analyzed (Participants) | 3
  Surgical Completers, baseline | 72.00 (4.58)
  Surgical Completers, week 12: number analyzed (Participants) | 3
  Surgical Completers, week 12 | 8.00 (2.08)

9. Primary Outcome: Subjective Sinonasal Symptoms on 10cm Visual Analogue Scale(VAS)
Description: Minimum Score: 0 Maximum Score: 100 A higher score indicates a worse outcome.
Time Frame: baseline to week 56
Population: Intention-to-treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 29
units on a scale
  Medicine Completers, baseline: number analyzed (Participants) | 7
  Medicine Completers, baseline | 64.3 (7.5)
  Medicine Completers, week 56: number analyzed (Participants) | 7
  Medicine Completers, week 56 | 35.0 (9.2)
  Surgical Completers, baseline: number analyzed (Participants) | 3
  Surgical Completers, baseline | 90.0 (5.8)
  Surgical Completers, week 12: number analyzed (Participants) | 3
  Surgical Completers, week 12 | 16.7 (6.7)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment | Control | Open Label
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/29
Other Adverse Events (participants affected / at risk) | 8/10 | 5/10 | 18/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=10) | Control (N=10) | Open Label (N=29)
Acute Sinusitis (General disorders) | 3 (3) | 4 (4) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 4 (4) | 3 (3) | 2 (2)
Swelling of Hands or Feet (General disorders) | 3 (3) | 0 (0) | 2 (2)
Slow, Fast or Irregular Heart Rate (Cardiac disorders) | 2 (2) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 6 (6) | 1 (1) | 8 (10)
Heartburn (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (6)
Lightheadedness (General disorders) | 5 (5) | 2 (2) | 2 (2)
Headache (General disorders) | 3 (3) | 2 (2) | 6 (6)
Fainting (General disorders) | 0 (0) | 0 (0) | 0 (0)
Blurred Vision (General disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (General disorders) | 3 (3) | 0 (0) | 3 (3)
Tiredness (General disorders) | 5 (5) | 2 (2) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Yellow Eyes or Skin (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No